CLINICAL TRIAL: NCT02384174
Title: Resistant Starch and Non-starch Polysaccharide (Dietary Fibre) Intake in Relation to the Structure and Metabolic Activities of the Colonic Microbiome in Older People
Brief Title: Resistant Starch and Non-starch Polysaccharide (Dietary Fibre) Intake and the Colonic Microbiome in Older People
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2014GA05
Record Dates: First submitted 2015-02-20; First posted 2015-03-10 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Aging
Keywords: Aging; Resistant starch; Dietary fibre; Immune system; Bacteria; older subjects
MeSH Terms: interventions — Resistant Starch; Dietary Fiber; arabinogalactan; guar gum; Pectins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resistant starch (RS) (Experimental): Resistant starch (RS3)
  Interventions: Dietary Supplement: Resistant starch
- Dietary fibre (Experimental): Dietary fibre (Arabinogalactan, gum guar, pectin)
  Interventions: Dietary Supplement: Dietary fibre (arabinogalactan, gum guar, pectin)

INTERVENTIONS:
Dietary Supplement: Resistant starch
  Arms: Resistant starch (RS)
Dietary Supplement: Dietary fibre (arabinogalactan, gum guar, pectin)
  Arms: Dietary fibre

SUMMARY:
The development of preventative nutritional strategies to promote healthy ageing is becoming increasingly important. Elevated thresholds for taste and smell, coupled with swallowing difficulties and masticatory dysfunction, often result in nutritionally imbalanced diets among the elderly. This can induce great changes in the composition and metabolic activities of the gut microbiome, leading to decreased intestinal motility and impaired bowel function. This can result in constipation or diarrhoea, increased basal levels of inflammation, immunosenescence and morbidity. The objectives of this study are to use dietary modification to improve gut health in older people. Diets high in resistant starch or dietary fibre will be given to 50 elderly volunteers (70-95 years) living in the community, in a randomised double-blind cross-over study. The aim is to investigate the effects on microbiome composition and functionality through fermentation, reduced putrefaction, and modification of blood markers associated with obesity and diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 70-95 years, with BMI 18.5-30.0 kg m2.

Exclusion Criteria:

* Exclusion criteria will include asplenia and other acquired or congenital immunodeficiencies
* Any autoimmune disease
* Self-reported symptoms of acute or recent infection (including use of antibiotics within the previous 3 months)
* Taking probiotics or prebiotics, including lactulose for constipation
* Chronic gastrointestinal problems (e.g. Inflammatory Bowel Disease, Irritable Bowel Syndrome, cancer).
* Specifically, volunteers who are diabetic will not be excluded from the investigation.
* Assessment will be on a case by case basis.

Ages: 70 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2017-01 (Estimated); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with change in levels of faecal bifidobacteria measured by quantitative fluorescent in situ hybridisation (FISH). | 4 weeks

SECONDARY OUTCOMES:
Number of participants with change in the bacterial composition of the faecal microbiome measured by quantitative FISH. | 4 weeks
Number of participants with change in inflammatory markers linked to ageing measured in whole blood by enzyme linked immunosorbent assay (ELISA). | 4 weeks
  Measurement of cytokines Interleukin 6 (IL-6), Tumour necrosis factor-alpha (TNF-alpha), IL-1, IL-10, Interferon-gamma (INF-gamma), IL-4, IL-8, Monocyte chemoattractant protein 1( MCP-1) and serum C-reactive protein (CRP).
Number of participants with change in faecal genotoxic potential determined by measurement of faecal bacterial enzymes involved in the formation of genotoxic metabolites in the gut. | 4 weeks
  Enzymes to be measured beta-glucosidase, beta-glucuronidase, azoreductase, nitroreductase
Number of participants with a change in bowel habit and quality of life measured by completion of a bowel habit diary and quality of life questionnaire. | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiovascular and Diabetes Medicine/Gastroenterology, Ninewells Hospital and Medical School, Dundee, Tayside, United Kingdom

REFERENCES:
- [Background] Woodmansey EJ, McMurdo ME, Macfarlane GT, Macfarlane S. Comparison of compositions and metabolic activities of fecal microbiotas in young adults and in antibiotic-treated and non-antibiotic-treated elderly subjects. Appl Environ Microbiol. 2004 Oct;70(10):6113-22. doi: 10.1128/AEM.70.10.6113-6122.2004. PMID 15466557
- [Background] Bartosch S, Fite A, Macfarlane GT, McMurdo ME. Characterization of bacterial communities in feces from healthy elderly volunteers and hospitalized elderly patients by using real-time PCR and effects of antibiotic treatment on the fecal microbiota. Appl Environ Microbiol. 2004 Jun;70(6):3575-81. doi: 10.1128/AEM.70.6.3575-3581.2004. PMID 15184159
- [Background] Macfarlane S, Cleary S, Bahrami B, Reynolds N, Macfarlane GT. Synbiotic consumption changes the metabolism and composition of the gut microbiota in older people and modifies inflammatory processes: a randomised, double-blind, placebo-controlled crossover study. Aliment Pharmacol Ther. 2013 Oct;38(7):804-16. doi: 10.1111/apt.12453. Epub 2013 Aug 20. PMID 23957631